CLINICAL TRIAL: NCT05817552
Title: Accuracy of CBCT Imaging and Intraoral Scanner in Dental Plaster Casts Digitization: A Validity and Reliability Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Sayed Badry, Principle Investigator, Cairo University
Other Study IDs: ORAD3-3-1
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Dental Cast Digitization
Keywords: CBCT - Intraoral scanner - Cast digitization

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CBCT: Casts STLs generated from CBCT planmeca Pro Max
  Interventions: Diagnostic Test: Geomagic Control X
- Intraoral Scanner: Casts STLs generated from intraoral scanner Haron from 3DISC
  Interventions: Diagnostic Test: Geomagic Control X
- Desktop Optical Scanner: Casts STLs generated from desktop optical scanner Medit T710
  Interventions: Diagnostic Test: Geomagic Control X

INTERVENTIONS:
Diagnostic Test: Geomagic Control X — 3D Surface matching and compare

SUMMARY:
The Objective of this study is to evaluate the accuracy of CBCT and intraoral scanner, in digitization of dental plaster casts, by comparing them to desktop optical scanner as a gold standard.

DETAILED DESCRIPTION:
The Objective of this study is to evaluate the accuracy of CBCT and intraoral scanner, in digitization of dental plaster casts, by comparing them to desktop optical scanner as a gold standard.

Planmeca CBCT Modality, Haron 3DISC intraoral scanner will be used as index tests, and Medit T710 desktop optical scanner will be used as the gold standard.

STL files from test scanning modalities will be compared using the surface matching software (Geomagic control X). The surface matching software will automatically register the two compared STL files together using the best-fit alignment tool and will generate the 3D compare for the surface comparison between them.

ELIGIBILITY:
Inclusion Criteria:

* Adult dental casts with complete dentition and/or partially edentulous regions.
* Maxillary and mandible casts are both included.
* Intact casts without voids, cracks, or visible porosities

Exclusion Criteria:

* Casts of pediatric patients.
* Completely edentulous casts.
* Casts with hypodontia, supernumerary teeth or fractured teeth.
* Casts with retainers, metallic appliances, or partial dentures.
* Casts with voids, fractures, cracks or visible porosities.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Dental Plaster Casts
Sampling Method: Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Trueness | 1 year
  Trueness of the CBCT and intraoral scanner to generate digital model compared to desktop optical scanner

SECONDARY OUTCOMES:
Precision | 1 year
  Precision of the CBCT and intraoral scanner to generate digital models

IPD SHARING:
Plan to Share IPD: No